CLINICAL TRIAL: NCT05452746
Title: Acupuncture Augmentation Therapy for In-hospital Patients With Major Depression Disorder: a Pragmatic, Randomized Controlled Trial
Brief Title: Acupuncture Augmentation for Inpatients With Major Depression Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Mental Health, Singapore (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMHSingapore
Record Dates: First submitted 2022-06-24; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Depression
Keywords: Acupuncture
MeSH Terms: conditions — Depression | interventions — Acupuncture Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized single blinded controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor blinded to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental)
  Interventions: Device: Acupuncture
- Treatment as usual (Active Comparator)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Device: Acupuncture — Unilateral and bilateral acupuncture points:
  Du 20 and GV 29,39 MS1, MS2, MS3 and MS4,40
  Location of points:
  Number of needles: 9
  Depth of insertion:
  MS1, MS2, MS3: insert the needle obliquely in the frontal direction for 1 cm Du 20: insert the needle obliquely in the frontal direction for 0.5 cm GV 29: insert the needle obliquely and downward for 0.5 cm Needles retained for 20 min Needle type: Han Yi 0.25x25 mm Treatment regimen: once per day for 2 weeks
  Arms: Acupuncture
Other: Treatment as usual — Inpatient psychiatric care for depression
  Arms: Treatment as usual

SUMMARY:
Acupuncture practice is based on Traditional Chinese Medicine (TCM) principles of harmonization and balance, and the need to maintain unobstructed flow of energy (Qi) to attain efficient body functioning and metabolism so as to attain good mental and physical state of health. While increasing numbers of patients are seeking acupuncture treatment for depression in recent years, there is limited evidence of the effectiveness of acupuncture for in-hospital patients with severe depressive conditions and comorbid cognitive dysfunction, who need intensive antidepression care.

In this study, we propose a randomized clinical trial to test the clinical efficacy of acupuncture treatment for in-hospital patients who are suffering from major depressive disorder. A total of 84 patients will be 1:1 randomly assigned to 1 of 2 groups in a single-blind randomized controlled trial. The specific intervention arm involved daily augmentation TCM-style acupuncture with manual stimulation for total 10 sessions; the control arm is consisted of patients with treatment as usual (TAU), i. e. waitlist condition who will receive standard antidepressant medication with or without psychotherapies. Patients in TAU arm will be offered one free course (total 10 sessions) of acupuncture treatment in TCM outpatient clinic after they have been discharged from the ward. All patients' depressive symptoms, cognitive function, quality of life and functioning will be assessed and compared at pre-treatment (baseline), immediately after in-hospital acupuncture treatment, one-month post-treatment and 3-month post-treatment. In addition, we will analyze the association of sociodemographic and clinical characteristics with the treatment effect of acupuncture.

This study will be the first study to examine whether acupuncture is a viable augmentation treatment for in-hospital patients with depression. Expected outcomes will include determining the relative short and medium-term clinical effects from the most commonly used acupuncture treatment modalities in a local and multiethnic population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years.
2. DSM-V diagnosis of current Major Depressive Episode.
3. Montgomery-Asberg Depression Rating Scale score of 20 or more.
4. Able to give informed consent.

Exclusion Criteria:

1. History of psychosis or mania
2. With current ECT or neurostimulation treatment.
3. With severe heart or renal condition
4. Currently taking blood thinning drug including Aspirin etc.
5. Endocrine abnormalities (e.g., hypothyroidism, unstable diabetes);
6. History of central nervous system involvement (e.g., seizures, brain injury, neurologic ill- ness);
7. Pregnancy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) (objective, clinician administered). | 2 week post treatment
  MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorder (scored 0 to 60 with higher scores meaning worse outcome)
Montgomery-Åsberg Depression Rating Scale (MADRS) (objective, clinician administered). | 1 month post treatment
  MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders.(scored 0 to 60 with higher scores meaning worse outcome)
Montgomery-Åsberg Depression Rating Scale (MADRS) (objective, clinician administered). | 3 months post treatment
  MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders.(scored 0 to 60 with higher scores meaning worse outcome)

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) (clinician administered). | 2 weeks, 1 month, 3 months post treatment
  MoCA was validated in the setting of mild cognitive impairment,44 and has subsequently been adopted in numerous other settings clinically. (scored 0 to 30 with higher scores indicating better outcome)
EQ-5D (self-administered) | 2 weeks, 1 month, 3 months post treatment
  EQ-5D is a standardized measure of health-related QoL developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys
Quick Inventory of Depressive Symptomatology- Self report 16 items (QIDS-SR16) (subjective, self-administered) | 2 weeks, 1 month, 3 months post treatment
  The QIDS-SR16 has highly acceptable psychometric properties, which supports the usefulness of this brief rating of depressive symptom severity in both clinical and research settings
Global Assessment of Functioning (GAF) (clinician administered) | 2 weeks, 1 month, 3 months post treatment
  GAF is a scoring system that mental health professionals use to assess how well an individual is functioning in their daily lives (Scored 0-100 with higher score indicating better outcomes)
TCM Assessment Form (Depression) | 2 weeks, 1 month, 3 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Phern Chern Tor, MBBS, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Institute of Mental Health, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No